CLINICAL TRIAL: NCT04779801
Title: Attachment-Based Family Therapy for Adolescents With Transdiagnostic Binge Eating
Brief Title: Attachment-Based Family Therapy for Adolescents With Binge Eating
Acronym: ABFT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Drexel University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004007768
Record Dates: First submitted 2021-02-25; First posted 2021-03-03 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2020-12

CONDITIONS: Bulimia Nervosa; Binge-Eating Disorder; Other Specified Feeding or Eating Disorder
MeSH Terms: conditions — Bulimia Nervosa; Binge-Eating Disorder; Feeding and Eating Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ABFT (Experimental): Adolescents and one or both parents will complete 16 weeks of Attachment-Based Family Therapy treatment.
  Interventions: Behavioral: Attachment-Based Family Therapy

INTERVENTIONS:
Behavioral: Attachment-Based Family Therapy — 16 weeks of Attachment-Based Family Therapy treatment.

SUMMARY:
The purpose of this study is to examine whether Attachment-Based Family Therapy (ABFT), a well-validated treatment for adolescents with depression and suicidality, is feasible and acceptable for adolescents with binge eating and their families.

DETAILED DESCRIPTION:
This study involves a phone screen and baseline assessment to determine eligibility. Participants who are eligible for the study will receive 16 weeks of ABFT treatment. The treatment primarily focuses on improving communication and relationships within the family, and will also address disordered eating behaviors (e.g., binge eating, laxative use, self-induced vomiting). All participants enrolled in the study will receive the same treatment. Participants will also complete research assessments throughout treatment, at the end of treatment, and 3-months after the end of treatment. Research assessments include a battery of questionnaires and interviews.

ELIGIBILITY:
Inclusion Criteria:

* Speak, write, and understand English
* Age 12-22 years old
* Have a diagnosis of DSM-5 AN, BN, BED, or OSFED
* Medically stable for outpatient treatment
* Must have a parent, guardian, or primary caregiver who is willing to participate in the study and treatment

Exclusion Criteria:

* Acute suicide risk
* No parent or guardian agreement to participate
* Are currently receiving psychological treatment for an eating disorder
* Are currently receiving weight loss treatment
* Co-morbid clinically significant psychological disorder that would require attention beyond the study treatment (e.g., psychotic disorder, substance dependence)
* Diagnosis of intellectual disability

Ages: 12 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-12-10 (Actual); Primary Completion 2021-12-10 (Estimated); Study Completion 2022-04-10 (Estimated)

PRIMARY OUTCOMES:
Five-Minute Speech Sample (FMSS) | Change in critical comments and emotional overinvolvement from baseline to treatment completion, at 16 weeks
  The Five-Minute Speech Sample is a widely-used interview to assess critical comments and emotional overinvolvement in families.

SECONDARY OUTCOMES:
Eating Disorder Examination (EDE) | Change in frequency of binge-eating and, if applicable, purging from baseline to treatment completion, at 16 weeks
  The Eating Disorder Examination is a widely-used, semi-structured interview for the assessment of eating disorder symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Drexel University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No